CLINICAL TRIAL: NCT01071239
Title: A Phase II Trial of Hematopoietic Stem Cell Transplantation for the Treatment of Patients With Fanconi Anemia Lacking a Genotypically Identical Donor, Using a Chemotherapy Only Cytoreduction With Busulfan, Cyclophosphamide and Fludarabine
Brief Title: Hematopoietic Stem Cell Transplant for Fanconi Anemia
Acronym: FA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, David A. Margolis, Professor of Pediatrics and BMT Program Director, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FA 08/89
Record Dates: First submitted 2009-05-20; First posted 2010-02-19 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Fanconi Anemia
Keywords: Fanconi Anemia; Hematopoietic stem cell transplant
MeSH Terms: conditions — Fanconi Anemia | interventions — Busulfan; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone marrow processing (Experimental): Bone Marrow processing using the CliniMACs device
  Interventions: Device: CliniMACs device; Drug: Busulfan; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: ATG

INTERVENTIONS:
Device: CliniMACs device — Donor Peripheral blood progenitor cells will use CD34+ selection with the use of the CliniMACs device
  Other Names: Milteny Biotec CliniMACS device
Drug: Busulfan — Chemotherapy administered as a part of the HSCT conditioning regimen.
Drug: Fludarabine — Chemotherapy administered as a part of the HSCT conditioning regimen.
Drug: Cyclophosphamide — Chemotherapy administered as a part of the HSCT conditioning regimen.
Drug: ATG — Chemotherapy administered as a part of the HSCT conditioning regimen.

SUMMARY:
The trial proposed is a single arm phase II treatment protocol designed to examine engraftment, toxicity, graft-versus-host disease, and ultimate disease-free survival following a novel cytoreductive regimen including busulfan, cyclophosphamide and fludarabine and anti-thymocyte globulin (ATG- a non-chemotherapy drug whose role is to kill your immune system) for the treatment of patients with Fanconi anemia who have severe aplastic anemia (SAA), or myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML), lacking HLA-genotypically identical donors using stem cell transplants derived from (1) HLA-compatible unrelated donors or (2) HLA haplotype-mismatched related donors.

DETAILED DESCRIPTION:
We are currently recruiting patients.

ELIGIBILITY:
Inclusion Criteria:

* Fanconi Anemia (confirmed by mitomycin C or DEB chromosomal breakage testing and one of the following hematological diagnoses: Severe Aplastic Anemia, Myelodysplastic Syndrome, Acute Myelogenous Leukemia
* Karnofsky or Lansy performance scale > or = to 70%.
* Must have adequate cardiac, hepatic, renal and pulmonary function.
* Must have 7/8 or 8/8 available unrelated donor.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Active CNS leukemic involvement
* Active uncontrolled viral, bacterial or fungal infection
* Positive for HIV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-04; Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
To measure the incidence and quality of engraftment and hematopoietic reconstitution. | 1, 3, 6 and 12 months post transplant date
  To measure the incidence and quality of engraftment and hematopoietic reconstitution.

SECONDARY OUTCOMES:
The incidence of early transplant related mortality and incidence and severity of acute and chronic GVHD | weekly for the first 30 days and then 3, 6, and 12 months post transplant date
  The incidence of early transplant related mortality and incidence and severity of acute and chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: David A Margolis, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States